CLINICAL TRIAL: NCT02567175
Title: Domperidone Expanded Access Protocol for Patients With Gastrointestinal Disorders
Status: No longer available | Type: Expanded Access
Sponsor: Prasanna K Kapavarapu (Other)
Responsible Party: Sponsor-Investigator, Prasanna K Kapavarapu, Attending Physician, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Other Study IDs: 14-010908
Record Dates: First submitted 2015-10-01; First posted 2015-10-02 (Estimated); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Gastroesophageal Reflux; Gastroparesis; Chronic Constipation With Overflow; Pseudo Obstruction
MeSH Terms: conditions — Gastroesophageal Reflux; Gastroparesis | interventions — Domperidone

INTERVENTIONS:
Drug: Domperidone
  Other Names: Motilium

SUMMARY:
FDA currently allows patients 12 years of age and older with various gastrointestinal (GI) conditions to be treated with Domperidone through the Expanded Access to Investigational Drugs program. These conditions include gastroesophageal reflux disease with upper GI symptoms, gastroparesis, and chronic constipation. Patients must have failed standard therapies to be eligible to receive Domperidone. This program facilitates availability of investigational drugs, (such as Domperidone) to patients with serious diseases or conditions when there is no comparable or satisfactory alternative therapy to diagnose, monitor, or treat the patient's disease or condition.

DETAILED DESCRIPTION:
Expanded Access Program Design:

The purpose of the Expanded Access Program is to provide oral Domperidone to patients' ≥12 years of age where, according to the investigator's judgment, a prokinetic effect is needed for the relief of refractory gastroesophageal reflux disease with upper gastrointestinal (GI) symptoms, gastroparesis, and chronic constipation.

The objective of the Expanded Access Program is to allow the use of Domperidone by patients with gastrointestinal disorders who have failed standard therapy. Failed standard therapy can be constituted by the following treatments: Proton Pump Inhibitor (PPI) Therapy, Erythromycin, allergy to medications. Subject must be on these therapies for a time period of 1 month before they are considered to be ineffective.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Age 12 and older
3. Symptoms or manifestations secondary to gastroesophageal reflux disease (GERD) (e.g., persistent esophagitis, heartburn, upper airway signs or symptoms or respiratory symptoms), gastrointestinal motility disorders such as nausea, vomiting, severe dyspepsia or severe chronic constipation that are refractory to standard therapy. Failed standard therapy can be constituted by the following treatments: PPI Therapy, Erythromycin, allergy to medications. Subject must be on these therapies for a time period of 1 month before they are considered to be ineffective.
4. Patients must have a comprehensive evaluation to eliminate other causes of their symptoms.
5. Patient or Parent/Legal Guardian has signed informed consent and child assent (as appropriate) for the administration of Domperidone that informs the patient of potential adverse events including:

   * increased prolactin levels
   * extrapyramidal side effects
   * breast changes
   * cardiac arrhythmias including QT prolongation and death
   * There is a potential for increased risk of adverse events with the drugs listed in the Domperidone protocol addendum (see Appendix).
6. Patients with a weight > 35kg
7. Patients are able to swallow the Domperidone pill.

Exclusion Criteria:

1. History of, or current, arrhythmias including ventricular tachycardia, ventricular fibrillation and Torsade des Pointes. Patients with minor forms of ectopy (PACs) are not necessarily excluded.
2. Clinically significant bradycardia, sinus node dysfunction, or heart block. Prolonged QTc (QTc> 450 milliseconds for males, QTc>470 milliseconds for females).
3. Hepatic dysfunction
4. Renal insufficiency
5. Clinically significant electrolyte disorders.
6. Gastrointestinal hemorrhage or obstruction
7. Presence of a prolactinoma (prolactin-releasing pituitary tumor).
8. Pregnant or breast feeding female
9. Known allergy to Domperidone
10. The use of medications that interact with Domperidone. a. Subjects may be required to stop use (wash-out) of medications that interact with Domperidone. If the subject is not willing or able to stop use of the interacting medication, they may be excluded or withdrawn from the study at the investigator's discretion. Based on the medication the subject may be required to stop-use or wash out from, the PI will determine the appropriate washout period using clinical judgment. Some medications may require much longer washout periods than others, and this will be explained to each respective subject that requires stopping a medication.

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States